CLINICAL TRIAL: NCT06229782
Title: Orbital Artery Doppler Ultrasound as an Ancillary Test for Diagnosing Brain Death: a Prospective, Single Blind Comparative Study
Brief Title: Orbital Artery Doppler Ultrasound in Brain Death
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korgün Ökmen (Other Government)
Responsible Party: Sponsor-Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Organization: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-15 /33
Record Dates: First submitted 2024-01-08; First posted 2024-01-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Brain Death
MeSH Terms: conditions — Brain Death | interventions — Ultrasonography, Doppler, Transcranial; Computed Tomography Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ODUS (Other): Orbital Doppler ultrasonography (ODUS)
  Patients in whom brain death was suspected and the diagnostic procedure was initiated underwent ODUS .ODUS were performed during the apnoea test and the first neurological examination. At the second neurological examination at 12 hours, ODUS were repeated.
  Interventions: Diagnostic Test: Orbital Doppler ultrasonography; Diagnostic Test: Transcranial Doppler ultrasonography; Diagnostic Test: Computed Tomography Angiography

INTERVENTIONS:
Diagnostic Test: Orbital Doppler ultrasonography — During measurement, Doppler settings were adjusted to detect low flow and the smallest available Doppler gate was used for all ODUS examinations. The imaging probe position for ODUS was used transversely and axially, and mean values were recorded. ODUS 10-18 MHz linear probe was used.
Diagnostic Test: Transcranial Doppler ultrasonography — During the measurement, Doppler settings were adjusted to detect low flow, and the minor available Doppler gate was used for all TDUS examinations. For TDUS, a temporal window was used approximately 1 cm above the midpoint of the line joining the lateral palpebral fissure and the external auditory meatus.
  Transcranial Doppler ultrasonography ( TDUS) 3-5 MHz convex array probe was used.
Diagnostic Test: Computed Tomography Angiography — Cranial Computed Tomography Angiography

SUMMARY:
Brain death is the irreversible loss of all activity in the brain, brainstem, and cerebellum, the part of the central nervous system that remains inside the skull.

The clinical diagnosis of brain death should be supported by ancillary tests that provide information about cerebral blood flow or electrical activity in the brain. Some of the ancillary tests that evaluate cerebral blood flow include transcranial Doppler ultrasonography (TDUS), computed tomography (CT) angiography (CTA), and catheter-based cerebral angiography.

This study hypothesized that Orbital Doppler ultrasonography (ODUS) alone is more effective than TDUS in detecting intracranial blood flow in diagnosing brain death. To this end, the investigators examined the results of ODUS in patients diagnosed as brain dead who underwent CT angiography.

ELIGIBILITY:
Inclusion Criteria:

* suspected brain death

Exclusion Criteria:

* eye surgery,
* uncontrolled diabetes mellitus,
* facial trauma,
* hypothermia,
* hypotension (systolic pressure < 100 mm Hg)
* endocrine-metabolic coma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-06-13 (Actual)

PRIMARY OUTCOMES:
ODUS | 30 minutes
  Orbital artery Doppler ultrasound (ODUS) ODUS measurements: T1; when brain death testing started; T2; 12 hours after the first measurement, T3; before CT angiography, T4; after CT angiography Peak systolic velocity (PSV) cm/s , end-diastolic velocity (EDV) cm/s measurement results. The absence of diastolic flow, reverse diastolic flow (oscillatory flow), and resistive index >1 were considered brain death.
Resistive index (RI) | 30 minutes
  The resistive index (RI) is a calculated flow parameter in ultrasound, derived from the maximum, minimum, and mean Doppler frequency shifts during a defined cardiac cycle. Along with the pulsatility index (PI), it is typically used to assess the resistance in a pulsatile vascular system.resistive index >1 were considered brain death.
  RI measurements: T1; when brain death testing started; T2; 12 hours after the first measurement, T3; before CT angiography, T4; after CT angiography .
  RI = (PSV - EDV) / PSV
  PSV = peak systolic velocity and EDV = end-diastolic velocity.

SECONDARY OUTCOMES:
Transcranial Doppler ultrasound (TDUS) | 30 minutes
  Transcranial Doppler ultrasound (TDUS) ultrasonography involves the use of a low-frequency (≤2 MHz) transducer, placed on the scalp, to insonate the basal cerebral arteries through relatively thin bone windows and to measure the cerebral blood flow velocity (CBFV) normal flow: mean = 55cm/sec. mild: > 120cm/sec. moderate: > 160cm/sec. s
Cerebral blood flow (CTA) | 40 minutes
  Transcranial Computed Tomography Angiography
Optic nerve diameter | 30 minutes
  Optic nerve diameter (mm) Orbital artery Doppler was performed simultaneously with ultrasound. The imaging probe position was used transversely and axially and mean values were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- University of Health Sciences,,Bursa Yuksek Ihtisas Training and Research Hospital,, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No